CLINICAL TRIAL: NCT02294981
Title: A Randomized Clinical Trial to Determine Whether a Novel Plaque-based Dosimetry Strategy Can Improve the Speed of Response to Treatment in Patients With Plaque Psoriasis (Photos)
Brief Title: Excimer Laser Phototherapy Outcomes in the Treatment of Psoriasis
Acronym: Photos
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol was changed to make it easier for treating doctors. No safety concerns
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14-15201
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Dosing (Active Comparator): Patients psoriasis to be treated with Excimer laser phototherapy based on conventional dosing guidelines. These guidelines determine the starting dose based on plaque thickness and the skin type of the patient. Patients will also be evaluated for psoriasis plaque response to test doses. The best dose will be selected from a test matrix of doses.
  Interventions: Device: Excimer laser phototherapy
- Plaque based dosing (Experimental): Patients will also be evaluated for psoriasis plaque response to test doses. The best dose will be selected from a test matrix of doses.
  Interventions: Device: Excimer laser phototherapy

INTERVENTIONS:
Device: Excimer laser phototherapy — Excimer laser phototherapy is a type of ultraviolet light that is applied to psoriatic plaques. It is administered using a laser in a targeted way so that only the plaques are treated (normal skin is not treated).

SUMMARY:
The purpose of this study is to determine the best dosing strategy when using Excimer Laser to treat plaque-type psoriasis. In this study, half of the body's psoriasis will be treated with a new dosing strategy, and the other half will be treated with the conventional method. We hope to show that the new dosing strategy will result in faster improvement of psoriasis.

DETAILED DESCRIPTION:
This is a randomized, assessor-blinded clinical trial to determine whether a novel plaque-based dosimetry strategy can improve the speed of response to excimer laser treatment in patients with plaque psoriasis. Each patient will receive plaque-based dosing on one side of the body and conventional dosing on the contralateral side. This design is based on the assumption that psoriasis usually affects patients in a symmetric distribution (e.g., knees and elbows) and the effect of excimer laser phototherapy is limited to the treated plaque. The side of the body treated with plaque-based dosimetry will be assigned using a table of random numbers. The assessor will be blinded to the treatment group. Each patient will be treated 1-2 times per week at the discretion of the investigator for a maximum of 10 treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic plaque psoriasis for at least 6 months
2. Age ≥ 18 years
3. Body surface area affected ≤ 10 percent
4. Presence of at least one pair of bilateral target lesions with an area of at least 20 cm2 per target lesion. The bilateral target lesions must be present in the same category of anatomical region (e.g., bilateral lower extremities, bilateral upper extremities or bilateral trunk).

Exclusion Criteria:

1. active or past history of erythrodermic psoriasis, guttate psoriasis, or pustular psoriasis
2. history of photosensitivity disorder
3. history of malignant melanoma
4. active, invasive non-melanoma skin carcinoma
5. Fitzpatrick Skin Type I
6. Subject has received ultraviolet B phototherapy or any topical anti-psoriatic therapy within two weeks prior to starting the study.
7. Subject has received systemic or topical psoralen-ultraviolet A photochemotherapy within four weeks prior to starting the study.
8. Subject has received biologic therapy within three months of starting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Bhutani, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis Skin and Treatment Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient lost to follow-up
Groups:
- Conventional Dosing/Plaque Based Dosing: Patients psoriasis to be treated with Excimer laser phototherapy based on conventional dosing guidelines. These guidelines determine the starting dose based on plaque thickness and the skin type of the patient. Patients will also be evaluated for psoriasis plaque response to test doses. The best dose will be selected from a test matrix of doses.
  Excimer laser phototherapy: Excimer laser phototherapy is a type of ultraviolet light that is applied to psoriatic plaques. It is administered using a laser in a targeted way so that only the plaques are treated (normal skin is not treated).
Period: Overall Study
Arm/Group | Conventional Dosing/Plaque Based Dosing
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Conventional Dosing/Plaque Based Dosing
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 45 [29 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Modified Psoriasis Area Severity Index
Description: The Modified Psoriasis Area Severity Index is a scale that grades psoriasis based on thickness, redness, scaling, and area involvement.
Time Frame: 10 weeks
Population: The sponsor decided to stop the current trial and start a new, larger multi center sponsored study. The results were not analyzed due to termination of study.
Arm/Group | Conventional Dosing/Plaque Based Dosing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reviewed at each participant visit (once or twice weekly) for the duration of the study (total of 5 months).
Description: No patients reported SAEs, no deaths occurred during this study, no AEs of any type was reported during this study.
Arm/Group | Conventional Dosing/Plaque Based Dosing
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The sponsor decided to stop the current trial and start a new, larger multi center sponsored study. The results were not analyzed due to termination of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02294981/Prot_SAP_000.pdf